CLINICAL TRIAL: NCT06377761
Title: A Randomized, Double-blind, Placebo-controlled Study on the Treatment of Heart Failure with Preserved Ejection Fraction with Qishen Granules Based on Cardiopulmonary Exercise Test
Brief Title: Study on Heart Failure with Preserved Ejection Fraction with Qishen Granules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lei Wang,MD, Chief Physician, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BF-2022-121
Record Dates: First submitted 2022-06-02; First posted 2024-04-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure with Preserved Ejection Fraction
Keywords: Heart Failure with Preserved Ejection Fraction; Qishen Granules; Cardiopulmonary Exercise Test

STUDY DESIGN:
Intervention Model Description: Random parallel grouping
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qishen Granules (Experimental): On the basis of standardized drug treatment for HFpEF, participants who met the inclusion criteria were randomly given Qishen Granule intervention on the day of inclusion, taking it twice a day for 90 days.
  Interventions: Drug: Qishen Granules
- Placebo (Placebo Comparator): On the basis of standardized drug treatment for HFpEF, participants who met the inclusion criteria were randomly given placebo granules on the day of inclusion, which were taken twice a day for 90 days (the placebo was basically the same as Qishen granules in terms of appearance, shape, color, taste, etc.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qishen Granules — One package per time, twice a day, 90 days of treatment
  Arms: Qishen Granules
Drug: Placebo — One package per time, twice a day, 90 days of treatment (the placebo was basically the same as Qishen granules in terms of appearance, shape, color, taste, etc.)
  Arms: Placebo

SUMMARY:
With the cardiopulmonary exercise testing as the primary outcome, the study aims to evaluate the efficacy of Qishen Granules on cardiac function, quality of life and biomarker level of patients with heart failure with preserved ejection fraction (HFpEF), which will provide evidence for the treatment of HFpEF with traditional Chinese medicine.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is common and is associated with high morbidity and mor-tality in China. Studies have shown that traditional Chinese medicine (TCM) combined with conventional Western medicine has a good effect on improving exercise tolerance and quality of life in patients with HFpEF, but there are still some shortcomings that limit the reliability and extrapolation of results. Based on TCM theory and our decades of experience, we developed Qishen Granules for therapeutic use in the treatment of HFpEF. The good effect of Qishen Granules in patients with heart failure has been clinically verified before. In this study, cardiopulmonary exercise test (CPET) was used to evaluate the peak oxygen consumption (peak VO2), which is the gold standard assessment of aerobic capacity. Therefore, we selected VO2 peak as the primary outcome. At the same time, we conducted a preliminary assessment of the efficacy of Qishen Granules in improving the quality of life in patients with HFpEF, using Kansas City Cardiomyopathy Questionnaire (KCCQ) as the secondary outcome, and combined with other CPET indicators, echocardiographic measures, NT-pro BNP level, growth STimulation expressed gene 2 (ST2), biomarkers of liver and kidney function, and TCM Four-Dimensional Diagnostic Information Scale (TCMFDIS) to objectively, accurately, and comprehensively evaluate the efficacy and safety of Qishen Granules in improving quality of life and exercise capacity in patients with HFpEF.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form
2. Age 18-85 years old
3. Heart failure was diagnosed ≥ 3 months before enrollment, The heart function classification II-IV of New York Heart Association (NYHA)
4. has ≥ 1 of the following: 1） Structural heart disease (left atrial enlargement and/or left ventricular hypertrophy) recorded by echocardiography at the time of enrollment；2）Hospitalization due to heart failure within 12 months before enrollment
5. Retention of ejection fraction: left ventricular ejection fraction (LVEF)≥50% (Echocardiography)
6. Increase of NTpro-BNP (patients without atrial fibrillation>220pg/mL, patients with atrial fibrillation>660pg/mL
7. If diuretics are being administered orally, the dose must be stable for ≥ 2 weeks before inclusion in the study
8. At the time of randomization, it was clinically stable without signs of decompensation of cardiac failure (judged by the investigator)

Exclusion Criteria:

1. Patients with decompensated heart failure
2. Glomerular filtration rate (eGFR)<30mL/min/1.73m 2
3. Atrial fibrillation or atrial flutter with obvious liver disease or ALT, AST 3 times higher than the upper limit of normal
4. Symptomatic hypotension or systolic blood pressure (SBP)<100mmHg at the time of inclusion or baseline
5. Resting heart rate recorded by echocardiography at the time of screening>110bpm
6. Currently participating in another research equipment or drug test, or less than 30 days after the completion of another research equipment or drug test or receiving other research treatment. Patients participating in purely observational trials will not be excluded
7. At present, people who are taking traditional Chinese medicine or Chinese patent medicine with similar effect to Qishen Granules
8. Be allergic to any component of Qishen granules (astragalus membranaceus, salvia miltiorrhiza, and black aconite)
9. Patients who refuse to sign the informed consent form or estimate poor compliance and women who are pregnant, nursing or planning to become pregnant during the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in peak oxygen uptake within the average minute (PeakVO2) compared to baseline on day 90 | At enrollment versus at day 90
  Measure the efficiency of peak oxygen intake by combining oxygen volume and time to report PeakVO2 in ml/min

SECONDARY OUTCOMES:
Changes in Mitral valve diastolic blood flow velocity (E) and Mitral annulus lateral and septal motion velocity (e') compared to baseline on day 90 | At enrollment versus at day 90
  Measure the blood flow velocity or motion velocity of specific areas in cm/s
Changes in E/e' ratio compared to baseline on day 90 | At enrollment versus at day 90
  E/e' ratio
Changes in Left Atrial Volume index (LAVI) compared to baseline on day 90 | At enrollment versus at day 90
  Left atrial volume (estimated from echocardiography measurement data) and body surface area (estimated based on height and weight) will be combined to report LAVI in ml/m^2
Changes in Left ventricular mass index (LVMI) compared to baseline on day 90 | At enrollment versus at day 90
  Left ventricle mass (estimated from echocardiography measurement data) and body surface area (estimated based on height and weight) will be combined to report LVMI in g/m^2
Changes in Score of Kansas City Cardiomyopathy Questionnaire (KCCQ) compared to baseline on day 90 | At enrollment versus at day 90
  Calculate the scores of the KCCQ questionnaire
Changes in blood N terminal pro B type natriuretic peptide(NT-proBNP) compared to baseline on day 90 | At enrollment versus at day 90
  Level of blood NT-proBNP in mmol/L
Changes in blood Growth STimulation expressed gene 2(ST2) compared to baseline on day 90 | At enrollment versus at day 90
  Level of blood ST2 in mmol/L
Changes in blood urea compared to baseline on day 90 | At enrollment versus at day 90
  Level of blood urea in mmol/L
Changes in blood creatinine compared to baseline on day 90 | At enrollment versus at day 90
  Level of blood creatinine in mmol/L

OTHER OUTCOMES:
Changes in Aspartate aminotransferase(AST) compared to baseline on day 90 | At enrollment versus at day 90
  Level of blood AST in mmol/L
Changes in Alanine aminotransferase(ALT) compared to baseline on day 90 | At enrollment versus at day 90
  Level of blood ALT in mmol/L
Number of participants with treatment-related adverse events | At enrollment versus at day 90
  Assess the incidence of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, doctorate, Study Director — Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, China
Locations (2):
- China (2):
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - WangLei, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Li Z, Su M, Song G, Guo S, Feng W, Chen W, Li C, Wang L, Wang W. Efficacy and safety of Qishen granule for treating heart failure with preserved ejection fraction: a study protocol for a multicenter, randomized, double-blind, placebo-controlled trial. BMC Complement Med Ther. 2025 Aug 6;25(1):298. doi: 10.1186/s12906-025-05029-z. PMID 40770799